CLINICAL TRIAL: NCT02869035
Title: Predicting Treatment Outcome in Major Depressive Disorder
Brief Title: Treatment Outcome in Major Depressive Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Center for Integrated Molecular Brain Imaging, Copenhagen, Denmak (Other); Psychiatric Centre Copenhagen (Unknown); Central Visitation, Region Hovedstaden (Unknown)
Responsible Party: Principal Investigator, Gitte Moos Knudsen, Chair, Professor, MD, DMSc, Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NP1
Record Dates: First submitted 2016-07-29; First posted 2016-08-16 (Estimated); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Major Depressive Disorder
Keywords: PET; Serotonin; 5-HT4R; MRI; fMRI; EEG; Cortisol awakening response; Oxidative stress; Mental health; Prediction of treatment response; Inflammation; 5-HTTLPR; Brain imaging; Early life stress; Selective Serotonin Reuptake Inhibitor; Escitalopram; Psychometrics; Moderate depression; Severe depression; ERP; rsfMRI; 11C-SB207145; Sexual function; MDD; Affective cognition; Cold cognition; Social cognition; Anxiety
MeSH Terms: conditions — Depressive Disorder, Major; Psychological Well-Being; Inflammation; Stress, Psychological; Depression; Anxiety Disorders | interventions — Escitalopram; Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treatment of MDD patients (Experimental): Treatment of MDD patients with escitalopram
  Interventions: Drug: Escitalopram
- Healthy controls (No Intervention): No treatment.
- Shift of treatment for MDD patients (Experimental): Treatment of MDD patients with duloxetine
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Escitalopram — Patients will be treated with an antidepressant drug (escitalopram) at flexible standard doses for 12 weeks. If no response after 4 weeks; shift to duloxetine arm.
  Arms: Treatment of MDD patients
Drug: Duloxetine — Patients who at 4 weeks of escitalopram have not responded will be shifted to duloxetine at flexible standard dosages.
  Arms: Shift of treatment for MDD patients

SUMMARY:
Major Depressive Disorder (MDD) is one of the most severe and frequently occurring brain disorders worldwide. It has been linked to serotonergic dysfunction, sexual dysfunction, vulnerability to stress and neuro-inflammation. However, at the same time the etiological understanding is limited. Most antidepressants act on the serotonin (5- HT) system, yet between 30-50 % of patients with MDD does not respond successfully to 5-HT acting drugs. Recent experimental models from our group suggest that cerebral 5-HT levels in vivo can be indexed through molecular brain imaging of the 5-HT 4 receptor (5-HT4R) with a novel Positron Emission Tomography (PET) ligand (11C-SB207145). Also, our human studies have confirmed that cerebral synaptic 5-HT is inversely related to 5-HT4R binding and this technique thus can be used to investigate the role of 5-HT tone in the brain in MDD with differential responses to standard antidepressant treatment. By using multimodal neuroimaging technology, we aim to determine the status of the 5-HT system prior to and after either successful or failed neuropharmacological intervention in a non-randomized longitudinal open clinical trial. 100 untreated patients with moderate to severe MDD will be included. Data collection from various neurobiological domains (i.e, 5-HT4R PET imaging, Magnetic Resonance Imaging (MRI), functional MRI (fMRI), electroencephalogram (EEG), psychometrics, neuropsychological tests, and peripheral biomarkers) will be conducted before, during and after 12 weeks of antidepressant treatment. The objective is to identify predictors of pharmacological antidepressant treatment response in depressed individuals before and after 8 weeks of antidepressant treatment.

DETAILED DESCRIPTION:
Study population and study program:

Patients will be recruited through a unique new central referral site for "depression packages" in The Mental Health Services in the Capital Region of Denmark. 100 patients with MDD, 18-65 years of age, with moderate to severe single or recurrent episode of MDD (Hamilton 17 item (HAMD-17) score > 17) will be recruited through this portal. All diagnoses will be confirmed by a specialist in psychiatry.

Before initiation of pharmacological antidepressant treatment with escitalopram, patients will receive baseline examinations as follows: 1) 5-HT4R imaging with 11C-SB207145 PET-scan, 2) EEG examinations, 3) structural MRI, 4) functional MRI , 5) neuropsychological testing, 6) peripheral markers of immune-active cell responses, oxidative stress, cortisol-levels, RNA, genotypes and epigenetic factors will be measured in urine, saliva and peripheral blood at baseline and across the study period. Repeated measures across the study period include: 7) psychometrics by using self-reported questionnaires covering trait and state, including mental distress related to depression and other psychopathology, 8) neuropsychological examinations as well as 9) clinical follow-up with interview based ratings of mental status.

Patients will be treated with escitalopram at flexible doses of 10-20 mg/day adjusted depending on effects and side effects, and participate in clinical follow-up sessions at week 1, 2, 4 and 8. Patients with no response to escitalopram after 4 weeks will be shifted to a secondary pharmacological treatment (duloxetine). A final visit to determine longer-term clinical outcome will be performed at week 12. Compliance, side-effects to antidepressant treatment, and depressive symptoms will be monitored at each follow-up session.

The Hamilton 6 items (HAMD-6) subscale has recently shown to be more sensitive to antidepressant response (Østergaard et al), and will be used to identify treatment response in patients. Patients with > 50 % reduction in HAMD-6 after 4 weeks will be defined as early responders, and those with additional < 5 points on the HAMD-6 scale after 8 weeks will be considered in remission. Patients with >25% response at week 4 and < 50% reduction in HAMD-6 after full intervention will be considered non-responders. The assessment program including brain imaging with PET 11C-SB207145 will be conducted before drug intervention is initiated and, depending on treatment outcome, again after 8 weeks of antidepressant treatment in 20 patients in remission (remitters) and 20 non-responding patients (non-responders).

UPDATE: As per April 3, 2017 the rescanned group has been expanded to include various response patterns in order to capture rescan data from patients on a spectrum from poor to excellent treatment response, since out of the first 17 included patients only 1 patient fulfilled the non-responder criterion defined above. Accordingly, the clinical outcome parameter in the context will be changes in HAM-D6 from baseline at week 8.

Healthy controls:

From previous studies conducted at the Neurobiological Research Unit, there is access to brain imaging data and baseline PET-SB207145 brain images among healthy controls as well as an associated biobank with stored blood specimens. During the trial, additional healthy controls will be included and will receive baseline examinations and repeated neuropsychological testing after 12 weeks.

Hypotheses:

1. 5-HT4R binding (as imaged by 11C-SB207145 PET) before treatment will predict antidepressant treatment outcome (remission vs non-response) in depressed patients; higher binding at baseline is hypothesized to be associated with a better treatment outcome. Likewise, secondary, 5-HT4R binding (as imaged by 11C-SB207145 PET) before treatment is expected to be associated with the magnitude of change from baseline in Hamilton score (HAMD-6) at 8 weeks.
2. Remitters will display a greater reduction in 5-HT4R binding (as imaged by 11C-SB207145 PET) after antidepressant treatment relative to non-responders.
3. Patients with MDD will have a higher 5-HT4R binding (as imaged by 11C-SB207145 PET) relative to healthy controls.
4. High amygdala reactivity in an "emotional faces" fMRI paradigm before treatment predicts remission in response to antidepressant treatment.
5. Amygdala response to exposure to negative emotional faces (fear and anger) and cerebral 5-HT4R binding is expected to be associated, both in cross-sectional comparison before treatment and with regard to longitudinal changes (changes from baseline).
6. In resting state fMRI (rsfMRI), we expect that changes from baseline in a functional network centered around dorsomedial prefrontal cortex and other networks centered around anterior cingulate cortex and posterior cingulate cortex (default mode network) respectively will predict treatment outcome.
7. Low activity in a brain network engaged in reward processing (as assessed by fMRI) will predict antidepressant treatment response (i.e. positive association between low activity and remitter- relative to non-responder group) both in cross-sectional comparison before treatment and with regard to longitudinal changes (changes from baseline).
8. We expect reduced evoked gamma-activity measured with EEG and "Event-related-potentials" (ERP) in MDD patients compared to controls.
9. Using EEG/ERP, we expect reduced alpha and theta cordance and higher theta band activity among remitters measured at baseline.
10. Higher levels of systemic inflammation will predict poor cognitive function at baseline, and a poor antidepressant treatment outcome.
11. A blunted cortisol awakening response (CAR) at baseline will predict a positive antidepressant treatment outcome.
12. Restored HPA-axis dynamics (increased CAR compared to baseline) at week 8 will be associated with a positive treatment outcome.
13. There will be a significant association between functional networks found by EEG and fMRI, both at baseline and as contrast between remitters and non-responders after 8 weeks.
14. Hippocampal volume will predict treatment outcome.
15. Patients with a low 5-HT4R binding (as imaged by 11C-SB207145 PET) at baseline before treatment will have a lower libido relative to patients with a high binding.
16. Patients who respond to antidepressant treatment with the most pronounced changes in 5-HT4R binding (as imaged by 11C-SB207145) will experience a larger degree of sexual side-effects; i.e., the magnitude of 5-HT4R binding changes from baseline will be positively associated with the degree of sexual side-effects.
17. Childhood abuse (defined by a composite measure of early life stress questionnaires) and anxious depression (defined as anxiety/somatization factor score in HAMD-17 > 7) predicts poor antidepressant treatment outcome.
18. We expect urinary markers of oxidatively generated DNA/RNA damage to increase more in responders than in non-responders.
19. With an exploratory approach it will be possible to identify a set of predictors of antidepressant treatment outcome. This explorative analysis includes genetics, epigenetics, peripheral and central neurobiological characteristics, neuropsychology testing outcomes, psychometry including self-reported mental distress, both cross-sectional at baseline and as longitudinal measures.

Ethical Aspects:

The study protocol complies with the Declaration of Helsinki II and approval by all relevant authorities will be obtained before initiation. All human volunteers will receive oral and written information about the given study and provide written informed consent before enrolment. The trial is monitored by a Good Clinical Practise unit for the relevant domains.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe depression
* Age 18-65 years
* No previous antidepressant treatment the last 2 months
* Informed and signed consent

Exclusion Criteria:

* More than one previous attempt with antidepressant drugs
* Duration of current depression more than 2 years
* Current or previous psychiatric severe co-morbidity
* Acute suicidal ideation
* Psychotic
* Previous non-response to Selective Serotonin Reuptake Inhibitor (SSRI)
* Contraindication for SSRI treatment
* More suitable with treatment of alternative anti-depressive drug.
* Severe somatic co-morbidity
* Somatic medicine that can influence the trial
* Contraindications for MR-scanning
* Previous exposure to radioactivity > 10 milli sievert (mSv) within the last year
* Alcohol or drug abuse
* Previous severe head trauma
* Pregnancy
* Breast-feeding
* Insufficient Danish skills

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-08; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Binary treatment outcome in terms of remission from depression. | Baseline to clinical follow-up at 8 weeks after antidepressant treatment.
  Treatment outcome defined as changes in HAMD-6 score after antidepressant treatment (remitters and non-responders as previously defined).
Baseline cerebral 5-HT4R binding as imaged by 11C-SB207145 PET. | Baseline.
  Latent variable construct of 5-HT4R level based on quantification of 5-HT4R binding in primary volumes of interest; neocortex, nucleus caudatus, putamen and hippocampus. Assessed in depressed patients and healthy controls.
Changes from baseline in cerebral 5-HT4R binding as imaged by 11C-SB207145 PET | Baseline to follow-up scan at 8 weeks after antidepressant treatment.
  Difference in latent variable construct of 5-HT4R level based on quantification of 5-HT4R binding in primary volumes of interest; neocortex, nucleus caudatus, putamen and hippocampus. Measured in remitters and non-responders.
Baseline hippocampus volume | Baseline.
  Structural MRI scan in depressed patients and healthy controls.
Changes from baseline in hippocampus volume. | Baseline to follow-up scan at 8 weeks after antidepressant treatment.
  Structural MRI in remitters and non-responders.
Baseline fMRI BOLD response to an emotional faces paradigm | Baseline
  fMRI (BOLD response) based assessment of brain activity to emotionally salient, relative to neutral, stimuli.
Changes from baseline in fMRI BOLD response to an emotional faces paradigm | Baseline to follow-up scan at 8 weeks after antidepressant treatment.
  fMRI (BOLD response) based assessment of brain activity to emotionally salient, relative to neutral, stimuli.
Baseline fMRI BOLD response to reward paradigm. | Baseline
  fMRI (BOLD response) based assessment of brain activity in response to reward, relative to non-reward, stimuli.
Changes from baseline in fMRI BOLD response to reward paradigm | Baseline to follow-up scan at 8 weeks after antidepressant treatment.
  fMRI (BOLD response) based assessment of brain activity in response to reward, relative to non-reward, stimuli.
Baseline rsfMRI based spontaneous co-fluctuations in low frequency BOLD signal (functional connectivity) | Baseline
  Assessed with rsfMRI scan in the resting state, i.e. non-goal oriented spontaneous thought and awake.
Changes from baseline in rsfMRI spontaneous co-fluctuations in low frequency BOLD signal (functional connectivity) | Baseline to follow-up scan at 8 weeks after antidepressant treatment.
  Assessed with rsfMRI scan in the resting state, i.e. non-goal oriented spontaneous thought and awake.
Sexual function in depression | Baseline
  Assessed with scores of self reported sexual function questionnaires in depressed patients and healthy controls.
Changes in sexual function | Baseline to clinical follow-up at 8 or 12 weeks after antidepressant treatment, and baseline to follow-up scan at 8 weeks after antidepressant treatment.
  Questionnaire-based self-reported sexual function in remitters and non-responders
Baseline EEG including event related potentials (ERP) | Baseline
  Assessment of evoked gamma activity, alpha and theta cordance band activity in depressed patients and healthy controls.
Changes in EEG including event related potentials (ERP) | Baseline to follow-up examination at 8 weeks after antidepressant treatment.
  Assessment of evoked gamma activity, alpha and theta cordance band activity in remitters and non-responders.
Cortisol awakening response | Baseline
  Cortisol changes in response to awakening as measured in saliva from 0 to 60 minutes after awakening in depressed patients and healthy controls.
Changes in cortisol awakening response (HPA-axis dynamics) | Baseline and follow-up examination at 8 weeks after antidepressant treatment.
  Measured in remitters and non-responders.
Systemic inflammation peripheral blood hsCRP and immunoactive cytokines | Baseline and follow-up examination at 8 weeks after antidepressant treatment.
  Measured with peripheral blood markers in plasma by high-sensitivity (hs) methods.
Changes in systemic inflammation peripheral blood hsCRP and immunoactive cytokines | Baseline and follow-up examination at 8 weeks after antidepressant treatment.
  Measured with peripheral blood markers in plasma by high-sensitivity (hs) methods.
Systemic oxidative stress in terms of 8-oxodG and 8-oxoGuo in urine | Baseline
  8-oxodG and 8-oxoGuo measured with mass spectrometry in spot-urine and normalized to urinary creatinine, in depressed patients and healthy controls.
Changes in systemic oxidative stress in terms of 8-oxodG and 8-oxoGuo in urine | Baseline and follow-up examinations at 8 weeks after antidepressant treatment.
  8-oxodG and 8-oxoGuo measured with mass spectrometry in spot-urine and normalized to urinary creatinine, in remitters and non-responders.
Early life Stress | Baseline
  Self-reported early life stress with the Children Abuse and Trauma Scale (CATS) questionnaire.
Performance on Verbal Affective Memory Tasks (VAMT-26). | From baseline to follow-up after 12 weeks of treatment with antidepressant treatment.
  Differences between healthy controls and depressed patients at baseline and week 12 follow-up, as well as longitudinal alterations to treatment response in MDD patients.
Performance on Moral Judgement Task | From baseline to follow-up after 12 weeks of treatment with antidepressant treatment.
  Differences between healthy controls and depressed patients at baseline and week 12 follow-up, as well as longitudinal alterations to treatment response in MDD patients.
Performance on Letter-Number Sequence Task. | From baseline to follow-up after 12 weeks of treatment with antidepressant treatment.
  Differences between healthy controls and depressed patients at baseline and week 12 follow-up, as well as longitudinal alterations to treatment response in MDD patients.

SECONDARY OUTCOMES:
Changes from baseline in HAMD-6 score | Baseline to follow-up at 8 and 12 weeks
  Score indexing changes in severity of the depressed state
HAMD-6 score after 8 and 12 weeks of antidepressant treatment | Week 8 and 12 of treatment period
  Score indexing severity of the depressed state
Regional 5-HT4R binding | Measured at baseline and after 8 weeks of antidepressant treatment.
  Measurement of 5-HT4R binding in (a) striatum (caudate nuclei and putamen), (b) a pooled limbic region (amygdala, hippocampus, thalamus, anterior- and posterior cingulate cortex,) (c) a pooled neocortex region (parietal cortex, occipital cortex, lateral temporal cortex, insula, orbito-frontal and lateral-frontal cortex).
Sexual side-effects from antidepressant treatment | 8 weeks of antidepressant treatment
  Perceived side effects from self reported questionnaires
Baseline latent variable construct of self-reported mental state | Baseline
  Composed by latent variable structural equation modelling of self-reported mental state from questionnaires score of: Becks Depression Inventory -II (BDI-II), Perceived Stress Scale (PSS), Snaith-Hamilton Pleasure Scale (SHAPS), Rumination Response Scale (RRS), Pittsburgh Sleep Quality Index (PSQI), Generalized Anxiety Distress Assessment 10 item (GAD-10), Activity level, Profile of Mood States (POMS), Visual Analogue Scale for mental distress (VAS) and Brief symptom Inventory-53 item (BSI-53)) in depressed patients and healthy controls.
Baseline self reported family history of mood disorders | Baseline
  Family History Assessment Module (OS-FHAM) in depressed patients and healthy controls.
Changes from baseline in self-reported mental state questionnaire-based latent variable construct | At baseline and repeated across the study period to last follow-up after 12 weeks of antidepressant treatment.
  Composed by latent variable structural equation modelling of changes from baseline in self-reported mental state from questionnaires score of: Becks Depression Inventory -II (BDI-II), Perceived Stress Scale (PSS), Snaith-Hamilton Pleasure Scale (SHAPS), Rumination Response Scale (RRS), Pittsburgh Sleep Quality Index (PSQI), Generalized Anxiety Distress Assessment 10 item (GAD-10), Activity level, Profile of Mood States (POMS) and Brief symptom Inventory-53 item (BSI-53) in remitters and non-responders.
Total daily cortisol output | Baseline (before treatment)
  Area under curve of 8 serial measures of salivary cortisol concentrations during an assessment day
Changes in total daily cortisol output | Baseline (before treatment) to 8 weeks of antidepressant treatment
  Difference in area under curve of 8 serial measures of salivary cortisol concentrations during an assessment day
Parental bonding quality | Baseline
  Self-reported parental bonding quality as assessed in baseline by parental bonding interview (PBI)
5-HTTLPR genotype status | Baseline
  5-HTTLPR genotype status (binary), i.e. high-expressing LALA vs low-expressing (S or LG) variants
Epigenetic FK506-binding protein 51 (FKBP5) status at baseline | Baseline
  Methylation of the FKBP5 gene
Changes in epigenetic FKBP5 status from baseline | Baseline to 8 and 12 weeks of intervention
  Changes in methylation status of the FKBP5 gene
Epigenetic 5-HTTLPR status at baseline | Baseline
  Methylation status of the 5-HTTLPR gene
Changes in epigenetic 5-HTTLPR status from baseline | Baseline to 8 and 12 weeks of intervention
  Changes in methylation status of the 5-HTTLPR gene
Epigenetic spindle and kinetochore associated complex subunit 2 (SKA2) status at baseline | Baseline to 8 and 12 weeks of intervention
  Methylation status of the SKA2 gene
Changes in epigenetic SKA2 status from baseline | Baseline to 8 and 12 weeks of intervention
  Changes in methylation status of the SKA2 gene
Performance on Face and Eyes Emotion Recognition Task | From baseline to follow-up after 12 weeks of treatment with antidepressant treatment.
  Differences between healthy controls and depressed patients at baseline and week 12 follow-up, as well as longitudinal alterations to treatment response in MDD patients.
Performance on Intensity Morphing Task | From baseline to follow-up after 12 weeks of treatment with antidepressant treatment.
  Differences between healthy controls and depressed patients at baseline and week 12 follow-up, as well as longitudinal alterations to treatment response in MDD patients.
Performance on Social Information Preference Task | From baseline to follow-up after 12 weeks of treatment with antidepressant treatment.
  Differences between healthy controls and depressed patients at baseline and week 12 follow-up, as well as longitudinal alterations to treatment response in MDD patients.
Performance on Simple Reaction Time. | From baseline to follow-up after 12 weeks of treatment with antidepressant treatment.
  Differences between healthy controls and depressed patients at baseline and week 12 follow-up, as well as longitudinal alterations to treatment response in MDD patients.

CONTACTS AND LOCATIONS:
Overall Officials: Gitte M Knudsen, MD,Prof., Principal Investigator — Neurobiology Research Unit
Locations (1):
- Neurobiology Research Unit, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Via database of Center for Integrated Molecular Brain Imaging (Knudsen et al 2016, NeuroImage) data will be available for neuroscience research community contingent on approval by scientific board.

REFERENCES:
- [Background] Ostergaard SD, Bech P, Miskowiak KW. Fewer study participants needed to demonstrate superior antidepressant efficacy when using the Hamilton melancholia subscale (HAM-D(6)) as outcome measure. J Affect Disord. 2016 Jan 15;190:842-845. doi: 10.1016/j.jad.2014.10.047. Epub 2014 Nov 7. PMID 25487682
- [Derived] Jensen KHR, Aarestrup MR, Larsen SV, Kohler-Forsberg K, Knudsen GM, Jorgensen MB, Frokjaer VG. Psychoneuroendocrine profiles of unmedicated men with major depressive disorder and associations to treatment effects and sexual side-effects. Neurosci Appl. 2024 Feb 23;3:104050. doi: 10.1016/j.nsa.2024.104050. eCollection 2024. PMID 40656082
- [Derived] Sankar A, Ozenne B, Dam VH, Svarer C, Jorgensen MB, Miskowiak KW, Frokjaer VG, Knudsen GM, Fisher PM. Association between brain serotonin 4 receptor binding and reactivity to emotional faces in depressed and healthy individuals. Transl Psychiatry. 2023 May 11;13(1):165. doi: 10.1038/s41398-023-02440-3. PMID 37169780
- [Derived] Ip CT, Ganz M, Ozenne B, Olbrich S, Beliveau V, Dam VH, Kohler-Forsberg K, Jorgensen MB, Frokjaer VG, Knudsen GM. Association between the loudness dependence of auditory evoked potential, serotonergic neurotransmission and treatment outcome in patients with depression. Eur Neuropsychopharmacol. 2023 May;70:32-44. doi: 10.1016/j.euroneuro.2023.02.008. Epub 2023 Feb 28. PMID 36863106
- [Derived] Weber S, Frokjaer VG, Armand S, Nielsen JH, Knudsen GM, Joergensen MB, Stenbaek DS, Giraldi A. Sexual function improves as depressive symptoms decrease during treatment with escitalopram: results of a naturalistic study of patients with major depressive disorder. J Sex Med. 2023 Feb 14;20(2):161-169. doi: 10.1093/jsxmed/qdac016. PMID 36763929
- [Derived] Dam VH, Stenbaek DS, Kohler-Forsberg K, Cheng Ip, Ozenne B, Sahakian BJ, Knudsen GM, Jorgensen MB, Frokjaer VG. Evaluating cognitive disturbances as treatment target and predictor of antidepressant action in major depressive disorder: A NeuroPharm study. Transl Psychiatry. 2022 Nov 8;12(1):468. doi: 10.1038/s41398-022-02240-1. PMID 36347845
- [Derived] Fisher PM, Ozenne B, Ganz M, Frokjaer VG, Dam VN, Penninx BW, Sankar A, Miskowiak K, Jensen PS, Knudsen GM, Jorgensen MB. Emotional faces processing in major depressive disorder and prediction of antidepressant treatment response: A NeuroPharm study. J Psychopharmacol. 2022 May;36(5):626-636. doi: 10.1177/02698811221089035. Epub 2022 May 13. PMID 35549538
- [Derived] Ip CT, Olbrich S, Ganz M, Ozenne B, Kohler-Forsberg K, Dam VH, Beniczky S, Jorgensen MB, Frokjaer VG, Sogaard B, Christensen SR, Knudsen GM. Pretreatment qEEG biomarkers for predicting pharmacological treatment outcome in major depressive disorder: Independent validation from the NeuroPharm study. Eur Neuropsychopharmacol. 2021 Aug;49:101-112. doi: 10.1016/j.euroneuro.2021.03.024. Epub 2021 Apr 25. PMID 33910154
- [Derived] Kohler-Forsberg K, Jorgensen A, Dam VH, Stenbaek DS, Fisher PM, Ip CT, Ganz M, Poulsen HE, Giraldi A, Ozenne B, Jorgensen MB, Knudsen GM, Frokjaer VG. Predicting Treatment Outcome in Major Depressive Disorder Using Serotonin 4 Receptor PET Brain Imaging, Functional MRI, Cognitive-, EEG-Based, and Peripheral Biomarkers: A NeuroPharm Open Label Clinical Trial Protocol. Front Psychiatry. 2020 Jul 23;11:641. doi: 10.3389/fpsyt.2020.00641. eCollection 2020. PMID 32792991